CLINICAL TRIAL: NCT03181022
Title: Development of an MI Implementation Intervention in Adolescent HIV Care Settings
Brief Title: The Tailored-Motivational Interviewing Project
Acronym: TMI Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Karen MacDonell, PhD, Associate Professor, Wayne State University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R34MH103049-01 (NIH)
Record Dates: First submitted 2017-05-25; First posted 2017-06-08 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: HIV
Keywords: Patient-Provider Communication; Motivational Interviewing; Medication Adherence
MeSH Terms: conditions — Medication Adherence | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase 1a (No Intervention): To develop a measure of MI fidelity to ensure methodological rigor, acceptability and feasibility of administration, and clinical usefulness (Phase 1a). Ratings of 200 recordings of full patient-provider interactions with ratings of thin slices (recording 1 minute every 5 minutes) will be compared.
- Phase 1b (No Intervention): To conduct evidence-based tailoring of MI training for adolescent HIV care settings (Phase 1b). Coding via sequential analysis will be conducted of the 200 recordings to identify those specific provider communication behaviors that predict subsequent youth motivational statements.
- Phase 2 (No Intervention): To collaboratively develop the implementation intervention with 2 clinic teams associated with the ATN (Phase 2). A formative evaluation will be done to provide local diagnostic data regarding barriers and facilitators to adoption and create development panels - local development teams made up of clinicians and administrators from the site, and study staff to address barriers and facilitators from formative evaluation and draft locally-customized clinical care and multi-level implementation strategies with initial sustainability plans.
- Phase 3 (Experimental): To pilot test the implementation intervention and process/outcome evaluation protocols at two ATN sites in preparation for a full-scale trial.
  Interventions: Behavioral: Motivational Interviewing

INTERVENTIONS:
Behavioral: Motivational Interviewing — HIV care providers will be asked to attend an MI training workshop lasting a total of 12 hours. The workshop will be conducted by members of the MI Network of Trainers. MI training relies on experiential activities and cooperative learning methods. After the training, study staff will monitor MI fidelity, or how providers are using the MI skills, using the MI Coach Rating Scale. This will occur 3 times prior to the training, 3 times during the practice period, and then quarterly. They will be asked to complete an audiotaped standardized patient interaction (approximately 30 minutes) with one of the study staff. These will be coded and providers will be informed of their competency level for all but the pre-training role plays. Coaching will be provided for all participants during the practice period. For the quarterly role plays, no coaching occurs unless their score indicates they need additional coaching (an additional 45 minute session with an MI trainer).
  Arms: Phase 3

SUMMARY:
The purpose of the Tailored Motivational Interviewing Project (TMI) is to develop an implementation intervention to increase evidence-based patient-provider communication strategies using a Motivational Interviewing (MI) framework.

DETAILED DESCRIPTION:
The goal of this implementation science study is to develop an implementation intervention to increase evidence-based patient-provider communication strategies using a Motivational Interviewing (MI) framework. Providers who demonstrate communication consistent with MI are informative, provide support and respect for the patient, and facilitate collaboration, and generally have patients who are more satisfied, more committed to treatment regimens, and have better health outcomes. MI is already embedded in the clinical guidelines for HIV care and HIV risk reduction. However, the inconsistent implementation of clinical guidelines is a constant concern. Fidelity of implementation refers to the degree to which staff members actually implement programs as intended by the developer, or how faithful they are to specification of the evidence-based practice. Several studies suggest that delivering MI with high fidelity can be difficult for many practitioners, but practitioners benefit from carefully designed, multicomponent interventions to help them understand and use evidence- based practices. These implementation interventions consist of a strategy or set of strategies to increase implementation of evidence-based practice. Thus, the primary goal of this study is to develop and pilot test a multi-level implementation intervention to increase MI fidelity and improve patient-provider communication in adolescent HIV care settings within the Adolescent Trials Network for HIV/AIDS (ATN). Leading the way in implementation science in health care is the VA's Quality Enhancement Research Initiative (QUERI), created to link research activities to clinical services in "real time" to promote the rapid uptake of best clinical practices and improvement in patient outcomes. Utilizing the QUERI model of implementation intervention development, this study will prepare for a full-scale implementation intervention trial with the following aims: 1) To develop a measure of MI fidelity to ensure methodological rigor, acceptability and feasibility of administration, and clinical usefulness (Phase 1a). This includes comparing ratings of 200 recordings of full patient-provider interactions with ratings of thin slices (recording 1 minute every 5 minutes); 2) To conduct evidence-based tailoring of MI training for adolescent HIV care settings (Phase 1b). Phase 1 also includes coding utilizing sequential analysis of the 200 recordings to identify those specific provider communication behaviors that predict subsequent youth motivational statements; 3) To collaboratively develop the implementation intervention with HIV clinic teams associated with the ATN (Phase 2). A formative evaluation will be conducted to provide local diagnostic data regarding barriers and facilitators to adoption and create development panels - local development teams made up of clinicians and administrators from the site, and study staff to address barriers and facilitators from formative evaluation and draft locally-customized clinical care and multi-level implementation strategies with initial sustainability plans; 4) To pilot test the implementation intervention and process/outcome evaluation protocols at two ATN sites (Phase 3) to prepare for a full-scale implementation trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients: HIV+, current patient in HIV adolescent care clinic
* Providers: Provider in HIV adolescent care clinic

Exclusion Criteria:

* Unable to consent to participate (lack of English fluency)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
MI Coach Rating Scale | Change from pre- to post-training and implementation (12 months)
  Fidelity to Motivational Interviewing by HIV care providers

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University Health Center, Detroit, Michigan
  - Adolescent AIDS Program, The Bronx, New York